CLINICAL TRIAL: NCT01475448
Title: Effects of Long Distance Running Training on the Posture and Movement Control of Sedentary Older Adults
Brief Title: Long Distance Running Training by Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Marcos Duarte, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FR-262790
Record Dates: First submitted 2011-11-03; First posted 2011-11-21 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2011-11

CONDITIONS: Physical Activity; Aging
Keywords: biomechanics; motor control; movement; walking; running; sedentarism; joint moment
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sedentary older adults - running (Experimental): Sedentary older adults (60 years old or more) recruited from local community
  Interventions: Other: Long distance training
- Sedentary older adults - walking (Active Comparator): Sedentary older adults (60 years old or more) recruited from local community
  Interventions: Other: Walking training

INTERVENTIONS:
Other: Long distance training — Long distance training during four months, 3 times per week
  Arms: Sedentary older adults - running
Other: Walking training — Walking training during four months, three times per week
  Arms: Sedentary older adults - walking

SUMMARY:
The goal of this project is to understand the effect of regular practice of long distance running on the posture and movement control of older adults.

For such, the investigators will conduct an experiment with longitudinal design where sedentary elderly individuals will be trained in long distance running for about 4 months.

DETAILED DESCRIPTION:
In a study the investigators conducted about elderly runners, the main observed difference by the first time was that elderly individuals present greater foot abduction (toe-out) during running than young adults. This alteration has been observed in elderly individuals in general during walking, and identified as a protective mechanism to not overload the medial compartment of the knee joint. It is also known that elderly individuals present a different joint torque distribution in the lower limbs during walking in comparison with young adults. However, it's not known the relation between the movement patterns, particularly the foot abduction pattern, and the mechanical load on the knee joint during running by elderly individuals and neither the longitudinal effect of running practice on this relation and on the mechanical joint load distribution. Another unknown aspect is the actual effect of the running practice on the posture control of elderly individuals.

With this project, the investigators want to understand why elderly individuals change their movement pattern during running, to determine for the same subjects if this altered pattern is also present during walking and standing, and to determine the effect of running practice on the elderly posture control. Our hypotheses are that the strategy of greater foot abduction is present in all movement tasks and that the use of this strategy is related to the integrity of the knee joint, even considering the highly active elderly individuals and that the practice of running contributes for a better postural control in this population.

These findings will contribute for a greater understanding of the benefits of the practice of running and the adaptations developed by the elderly runners and in this way to contribute for the prescription of this activity to the elderly population.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary
* Independent bipedal locomotion

Exclusion Criteria:

* Inapt for practicing physical activity
* Severe alteration of the muscle-skeletal system
* Cognitive or neurological deficit
* Use of orthosis for locomotion

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline of posture and movement patterns at 16 weeks | Two weeks before and two weeks after the training for sixteen months
  biomechanical and physiological measures of the posture and movement patterns

SECONDARY OUTCOMES:
Change from baseline of mechanical joint moments estimated by inverse dynamics at 16 weeks | Two weeks before and two weeks after the training for four months
  Estimated joint moments by inverse dynamics at the ankle, knee, and hip joints during the support phase of walking and running
Change from baseline of muscle activity measured by surface electromyography of selected muscles of the lower limb at 16 weeks | Two weeks before and two weeks after the training for four months
  Electromyographic activity of lower limb muscles during walking and running
Change from baseline of body sway measured by estabilography with a force plate during standing at 16 weeks | Two weeks before and two weeks after the training for four months
  Measurements of balance control during quiet and unconstrained standing using a force platform.

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Duarte, Principal Investigator — Federal University of ABC
Locations (1):
- Laboratory of Biophysics, São Paulo, São Paulo, Brazil